CLINICAL TRIAL: NCT00063505
Title: Genes of Hypertension in African Americans
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Theodore Kotchen, MD, Professor, Asssociate Dean for Clinical Research, Medical College of Wisconsin
Other Study IDs: 1216; R01HL070111 (NIH)
Record Dates: First submitted 2003-06-30; First posted 2003-07-01 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood cells and DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
To identify genes contributing to hypertension in African Americans by focusing on the physiological pathways that determine arterial pressure.

DETAILED DESCRIPTION:
BACKGROUND:

Since the mid 1990s, the investigators have extensively characterized African Americans for phenotypes related to cardiovascular and renal function. Based on recently completed genome scans, they have identified several chromosomal regions likely to contain genes influencing hypertension-related phenotypes in hypertensive, African American sib pairs. For several phenotypes, overlapping QTLs have also been identified in related studies in a genetically isolated French Canadian population and/or in homologous chromosomal regions in the F2 cross of Dahl-salt sensitive x normotensive Brown Norway rats.

DESIGN NARRATIVE:

The investigators will extensively phenotype 500 hypertensive and 500 normotensive African American subjects to conduct a genetic association study, using a single nucleotide polymorphism (SNP) genomic scan approach. To achieve a clear separation of blood pressures from hypertensive subjects, normotensive subjects will be selected from the lower third of the population-based blood pressure distribution. Hypertensive (BMI), and age. Inclusion of phenotypes is based on their relevance to the pathophysiology of hypertension and prior evidence of "heritability." Candidate genes for SNP analysis will be selected within chromosomal regions of two quantitative trait loci (QTLs) that they have previously demonstrated to be linked to hypertension-related phenotypes--a QTL for body mass index on chromosome 1 and a QTL for microalbuminuria on chromosome 18. SNP analyses will be carried out in 15 percent of the genes within each of these QTLs, and genes will be selected on the basis of their relevance to hypertension, including documented sequence conservation for blood pressure related QTLs with rat or mouse. The final goal of the project is to determine if distinct clusters of blood pressure related phenotypes can be identified that will permit stratification of hypertensive individuals into distinct subgroups to facilitate the analysis of the genetic determinants of hypertension and/or provide mechanistic leads to genes contributing to these traits.

ELIGIBILITY:
African Americans, age 18-75 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African Americans
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2002-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
genes of hypertension in African Americans | One time data collection
  There is no intervention

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Kotchen, Principal Investigator — Medical College of Wisconsin

REFERENCES:
- [Background] Grim CE, Cowley AW Jr, Hamet P, Gaudet D, Kaldunski ML, Kotchen JM, Krishnaswami S, Pausova Z, Roman R, Tremblay J, Kotchen TA. Hyperaldosteronism and hypertension: ethnic differences. Hypertension. 2005 Apr;45(4):766-72. doi: 10.1161/01.HYP.0000154364.00763.d5. Epub 2005 Feb 7. PMID 15699471